CLINICAL TRIAL: NCT04596462
Title: Characterizing Synovitis, Acne, Pustulosis, Hyperostosis, and Osteitis (SAPHO) With 68Ga-FAPI PET/CT
Brief Title: Characterizing SAPHO With 68Ga-FAPI PET/CT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHFAPISAPHO
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: SAPHO Syndrome
MeSH Terms: conditions — Acquired Hyperostosis Syndrome | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI PET/CT (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan.
  Interventions: Drug: 68Ga-FAPI

INTERVENTIONS:
Drug: 68Ga-FAPI — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image lesions of SAPHO by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitors

SUMMARY:
68Ga-FAPI has been developed as a tumor-targeting agent as fibroblast activation protein is overexpressed in cancer-associated fibroblasts and some inflammation. Thus this prospective study is going to investigate whether 68Ga-FAPI PET/CT may be superior for diagnosis, therapy response assessment and follow-up of SAPHO than 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Synovitis, acne, pustulosis, hyperostosis, and osteitis (SAPHO) syndrome is a spectrum of heterogeneous diseases characterized by osteoarticular and dermatological manifestations. Inflammatory osteitis with hyperostosis is the central feature of the syndrome, typically affecting multiple areas and possibly progressing to irreversible osteoarticular damage. Owing to the relapsing-remitting disease course, the goal of management is to improve clinical symptoms and prevent disease progression. Therefore, it's meaningful to seek appropriate methods to evaluate current osteroarticular lesions. 68Ga-FAPI that targets fibroblast activation protein (FAP) is introduced in tumor imaging. However, FAP was also shown to be expressed in rheumatoid arthritis, bone lesions with acute to chronic inflammation, fibrosis and ischemic heart tissue after myocardial infarction, thus the investigators speculate that it is possible for SAPHO to be imaged with 68Ga-FAPI. The aim of this study is to evaluate the performance of 68Ga-FAPI PET/CT in SAPHO and to compare it with the performance of 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed untreated SAPHO patients;
* 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against FAPI
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-FAPI PET/CT for SAPHO in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Metabolic parameters | through study completion, an average of 1 year
  Total Lesion Glycolysis (TLG) of SAPHO lesions are measured on 68Ga-FAPI PET/CT.
FAPI expression and SUV | through study completion, an average of 1 year
  Correlation between FAPI expression and SUV in PET
Disease burden assessement | through study completion, an average of 1 year
  Correlation between Total Lesion Glycolysis (TLG) of bone lesions assessed on 68Ga-FAPI PET/CT and clinical parameters for SAPHO

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Jing, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Dongcheng, China

IPD SHARING:
Plan to Share IPD: No